CLINICAL TRIAL: NCT01446822
Title: Transurethral Resection of Bladder Tumors Without Obturator Nerve Block or Relaxation: Extent of Adductor Muscle Contraction With Monopolar Versus Bipolar Resection Technique
Brief Title: Safety Study of Bipolar Versus Monopolar Transurethral Resection of Bladder Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Stephan Engeler (Other)
Responsible Party: Sponsor-Investigator, Daniel Stephan Engeler, Leitender Arzt, Klinik für Urologie, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URO-OBT-01
Record Dates: First submitted 2011-10-03; First posted 2011-10-05 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Neoplasm of Lateral Wall of Urinary Bladder
Keywords: urinary bladder neoplasm; bipolar transurethral resection; monopolar transurethral resection; obturator nerve
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bipolar transurethral resection (Experimental)
  Interventions: Device: Bipolar transurethral resection of the urinary bladder (PlasmaKinetic, Gyrus, Fresenius)
- Monopolar transurethral resection (Active Comparator)
  Interventions: Device: Monopolar transurethral resection of the urinary bladder (Storz GmbH &Co., Erbotom, Purisole)

INTERVENTIONS:
Device: Bipolar transurethral resection of the urinary bladder (PlasmaKinetic, Gyrus, Fresenius) — Lateral wall urinary bladder tumors are resected transurethrally without obturator nerve block or relaxation under general anesthesia. If resection not possible because of adductor muscle contraction, patients undergo relaxation.
  Other Names: PlasmaKinetic resectoscope; Gyrus PlasmaKinetic SuperPulse generator (Gyrus Medical Inc., Maple Grove, USA); Fresenius Natriumchlorid 9,0g/l (Fresenius Kabi AG, Homburg, Germany)
  Arms: Bipolar transurethral resection
Device: Monopolar transurethral resection of the urinary bladder (Storz GmbH &Co., Erbotom, Purisole) — Lateral wall urinary bladder tumors are resected transurethrally without obturator nerve block or relaxation under general anesthesia. If resection is not possible because of adductor muscle contraction, patients are treated by bipolar resection. If this is still not possible, they undergo relaxation.
  Other Names: Resectoscope Model 27050 (Karl Storz GmbH & Co. KG, Tuttlingen, Germany); Erbotom ICC 350 (Deltamed-ERBE AG,Winterthur, Switzerland); Purisole®SM (Fresenius Kabi AG, Homburg, Germany)
  Arms: Monopolar transurethral resection

SUMMARY:
This is a single-center, prospective, randomized, controlled trial comparing two established transurethral electrical resection methods of urinary bladder tumors regarding their risk of stimulating the obturator nerve.

One of the major safety issues with transurethral resection is bladder perforation as a consequence of obturator nerve stimulation followed by muscle contraction of. This is mostly a risk of resection of lateral bladder wall tumors near the course of the obturator nerve. It has been advocated that bipolar may be superior to monopolar resection, based on its different electrical properties. This is an important safety aspect for the patient.

Main study question: In patients with lateral wall urinary bladder tumors, is bipolar superior to monopolar transurethral electroresection regarding risk of stimulation of the obturator nerve without preoperative nerve block?

ELIGIBILITY:
Inclusion Criteria:

* neoplasms of the lateral wall of the urinary bladder (laterally to the corresponding ostium)
* operability given based on general medical condition
* informed consent

Exclusion Criteria:

* antiplatelet drugs stopped <7days (except acetylsalicylate <= 100mg p.o. qd)
* prothrombine time <70%
* age <18 years
* patronized Patients
* pregnancy
* severe poor medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Successful resection of bladder tumor | Intraoperative
  Successful resection of the neoplasm without relevant stimulation of the obturator nerve and consecutive contraction of the ipsilateral adductor muscles

SECONDARY OUTCOMES:
Complications | 3 months
  Degree of severity of the complications (perforation of the bladder, intraoperative bleeding, postoperative bleeding, others) according to the Clavien-classification

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Engeler, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital of St.Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Result] Gramann T, Schwab C, Zumstein V, Betschart P, Meier M, Schmid HP, Engeler DS. Transurethral resection of bladder cancer on the lateral bladder wall without obturator nerve block: extent of adductor spasms using the monopolar versus bipolar technique-a prospective randomised study. World J Urol. 2018 Jul;36(7):1085-1091. doi: 10.1007/s00345-018-2248-0. Epub 2018 Mar 1. PMID 29497859
- See also: Full text view of publication in World Journal of Urology — http://rdcu.be/H7MJ